CLINICAL TRIAL: NCT03766919
Title: Safety and Electrical Performance Evaluation of INVICTA Leads Models Equipped With DF4 Connector
Acronym: FRIENDS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: MicroPort CRM (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LNC001; CIV-PT-18-08-025366 (Other: INFARMED (Eudamed code))
Record Dates: First submitted 2018-10-16; First posted 2018-12-06 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Ventricular Arrythmia; Lead; ICD; Heart Failure
Keywords: INVICTA; Lead; ICD; CRT-D; MicroPort
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- INVICTA lead (Experimental): All patients eligible for enrolment in whom the INVICTA lead is attempted (Implant of the INVICTA lead)
  Interventions: Device: Implant of the INVICTA lead

INTERVENTIONS:
Device: Implant of the INVICTA lead — The implant or the attempt to implant an INVICTA lead

SUMMARY:
The primary objective of this study is to assess the safety and key electrical performance of the INVICTA leads equipped with DF4 connector: ACTIVE fixation type models (single and dual coil: INVICTA 1CR, INVICTA 2CR) and PASSIVE fixation type models (single and dual coil: INVICTA 1CT, INVICTA 2CT).

DETAILED DESCRIPTION:
FRIENDS study is a pre-market approval (INVICTA leads - devices under investigation - are not CE marked), interventional, prospective, longitudinal, international (European), multicenter, single arm study.

The devices under investigation, the INVICTA defibrillation leads, are new quadripolar leads, to be used with Implantable Cardiac Defibrillators and Cardiac Resynchronization Therapy Defibrillators (ICD/CRT-D).

This clinical study intends to demonstrate safety and electrical performances of the INVICTA leads among the different models: active fixation either single coil (model 1CR) or dual coil (model 2CR) and passive fixation, either single coil (model 1CT) or dual coil (model 2CT) leads models. The clinical data will be used to support the application to CE marking of INVICTA leads.

The primary endpoints will be evaluated at 3 months post-implantation; secondary endpoints will be evaluated up to 2 years post-implantation.

A maximum number of 224 patients will be enrolled in the study, in up to 60 centers in Europe.

The follow-up visits are scheduled at hospital discharge, at 1 month, at 3 months, at 6 months, at 12 months, at 18 months and at 24 months, post-implant .

ELIGIBILITY:
Inclusion Criteria:

1. Any patient presenting an ICD or CRT-D indication as detailed in the latest European Society of Cardiology (ESC) guidelines
2. Scheduled for a primary implant of an ICD / CRT-D, manufactured by MicroPort CRM and equipped with a RV DF4 connector
3. Signed and dated informed consent

Exclusion Criteria:

1. Tricuspid valvular disease or tricuspid replacement heart valve (mechanical or tissue)
2. Transient tachyarrhythmias due to reversible causes (such as drug intoxication, electrolyte imbalance, sepsis, hypoxia or other factors as myocardial infarction or electric shock)
3. Contraindication to a maximum single dose of 330 µg dexamethasone sodium phosphate (DSP)
4. Active myocarditis
5. Already included in another clinical study that could confound the results of this study
6. Inability to understand the purpose of the study or to meet follow-up visits at the implanting centre as defined in the investigational plan
7. Patient less than 18 years old or under guardianship or kept in detention
8. Known pregnancy, women in breastfeeding or in childbearing age without an adequate contraceptive method
9. Drug addiction or abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-12-27 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Freedom from INVICTA lead-related complications | 90 days
  Freedom from INVICTA lead-related complications as assessed by an independent events adjudicator and defined as any INVICTA lead-related serious adverse device effect (SADE) that resulted in patient death or required an additional invasive intervention.
INVICTA lead electrical performance at 3 months | 3 months
  Right Ventricular (RV) pacing threshold (V) of the INVICTA lead, measured by the implanted ICD/CRT-D with 0.5 ms pulse width

SECONDARY OUTCOMES:
INVICTA lead pacing threshold | 24 months
  RV lead pacing threshold amplitude (V), measured by the implanted ICD/CRT-D with 0.5 ms pulse width
INVICTA lead impedances | 24 months
  RV lead pacing impedance (Ohm) and defibrillation coil impedance (Ohm), measured by the implanted ICD/CRT-D
INVICTA sensing threshold | 24 months
  RV lead endocardial R wave amplitude (mV), measured by the implanted ICD/CRT-D
Percentage of the shocks that successfully terminate a ventricular arrhythmia episode | 24 months
  Percentage of endocardial shock therapies that successfully terminate ventricular arrhythmia episodes, calculated as the proportion of successful shocks on the total number of shocks delivered during defibrillation testing or spontaneous ventricular arrhythmias.
INVICTA lead complication free-rate up to 24 months | 24 months
  Report of INVICTA lead complication free-rate (complication defined as any INVICTA lead-related serious adverse device effect (SADE) that resulted in patient death or required an additional invasive intervention) up to 24 months post-implantation
INVICTA lead-related Serious Adverse Events and device deficiencies up to 24 months | 24 months
  Report of INVICTA lead-related SADEs and device deficiencies occurred up to 24 months post-implantation
INVICTA lead handling assessment | At Implant (Day 0)
  Summary of the investigators' opinion about INVICTA handling at implant
INVICTA lead implant success rate | At Implant (Day 0)
  % of enrolled patients successfully implanted with an INVICTA lead

CONTACTS AND LOCATIONS:
Overall Officials: Pedro MARQUES, MD, Principal Investigator — Hospital de Santa Maria - Lisboa - Portugal
Locations (10):
- France (3):
  - CHU, Brest
  - CHU, Clermont-Ferrand
  - CH de Valence, Valence
- Italy (2):
  - Cliniche Humanitas Gavazzeni, Bergamo
  - Ospedale Piemonte (IRCCS Bonino Pulejo), Messina
- Centro Hospitalar de Lisboa Norte - Santa Maria, Lisbon, Portugal
- Spain (4):
  - Hospital de Bellvitge, Barcelona, Hospitalet de Llobregat
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitari de Girona Doctor Josepj Trueta, Girona
  - Hospital Virgen de la Victoria, Málaga

IPD SHARING:
Plan to Share IPD: No